CLINICAL TRIAL: NCT02982096
Title: Randomized Controlled Pilot Study Comparing Healing With Epidermal Fractional Blistergrafting (CellutomeTM) to Acellular Technique (Membrane or Cream Dressings) in Superficial to Mid-dermal Burn Wounds
Brief Title: Study Comparing Healing With Epidermal Fractional Blistergrafting (CellutomeTM) to Acellular Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00003893
Record Dates: First submitted 2016-11-07; First posted 2016-12-05 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2021-09

CONDITIONS: Burn Wound
MeSH Terms: conditions — Burns | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cellutome treatment (Active Comparator): Cellutome Device: Use of Cellutome on burn wounds
  Interventions: Device: Cellutome Device
- Standard of Care (Other): Standard of Care: Acellular wound management
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Cellutome Device — Use of FDA approved Cellutome treatment on burn wounds
  Arms: Cellutome treatment
Other: Standard of Care — Acellular burn wound management
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine if healing occurs within 21 days of treatment with the use of the CellutomeTM device for fractional epidermal micro grafting compared with standard acellular techniques (creams and membrane dressings).

Healing will be determined by time to ≥90% epithelialization within 21 days of treatment. Cosmesis (as assessed by Vancouver Scar Scale (VSS), Patient Observer Scar Assessment Scale (POSAS), erythema, pigmentation, elasticity, thickness, and sensation) will be compared to standard techniques without application of skin cells (epidermal grafts = acellular) and will be measured twelve months post treatment application, ± 6 months.

DETAILED DESCRIPTION:
Hypothesis:

The use of epidermal blister grafting by the CellutomeTM device in the treatment of superficial and mid-dermal burn wounds will demonstrate a difference in time to healing compared to burn wounds treated with standard acellular technique.

Primary objective:

Determine if the use of the CellutomeTM device will demonstrate a difference in healing time compared to standard acellular technique. Final cosmetic outcomes (as assessed by Vancouver Scar Scale (VSS), Patient Observer Scar Assessment Scale (POSAS), erythema, pigmentation, elasticity, thickness, and sensation) will be assessed and described at 12 months ± 6 months post treatment.

Secondary objectives:

* Determine if donor sites have any visible scarring with the use of the CellutomeTM.
* Determine acute outcomes of therapy such as time to healing as assessed by ≥90% epithelialization.
* Determine chronic outcomes of therapy (as assessed by Vancouver Scar Scale (VSS), Patient Observer Scar Assessment Scale (POSAS), erythema, pigmentation, elasticity, thickness, and sensation).

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted or seen by the LVHN Burn Service with superficial to mid-dermal thickness burns will be considered for the study.
2. Age ≥18 years old.
3. Patients with a total body surface area (TBSA) burn > 1% outside of the face, neck, feet or genitalia, where at least 2 areas are greater in size than 5x5cm2 or at least one area that is greater than 10cm2

Exclusion Criteria:

1. Pregnant.
2. Age < 18 years old.
3. Proposed study area on face, neck, genitalia, or feet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Healing time comparison of the donor site wound at 12 months post baseline. | 12 months
  Assessed by Vancouver Scar Scale (Vascularity 0-3; Pigmentation 0-3; Pliability 0-5; and Height 0-4)
Healing time comparison of the donor site wound at 12 months post baseline. | 12 Months
  Assessed by Patient Observer Scar Assessment Scale (POSAS - evaluating patient perception of the scar including pain; itching; color; stiffness; thickness; irregularity on a 1-10 Likert Scale)
Healing time comparison of the donor site wound at 12 months post baseline. | 12 Months
  Visual assessment of Erythema of the donor site as compared to healthy skin
Healing time comparison of the donor site wound at 12 months post baseline. | 12 Months
  Assessed by measuring Elasticity (measured with cutometer) compared to healthy skin.
Healing time comparison of the donor site wound at 12 months post baseline | 12 Months
  Visual assessment of Pigmentation of the donor site as compared to healthy skin
Healing time comparison of the donor site wound at 12 months post baseline. | 12 Months
  Thickness of donor site (measured by ultrasound) compared to healthy skin
Healing time comparison of the donor site wound at 12 months post baseline. | 12 Months
  Sensation of donor site (measured by the Semmes-Weinstein filament tool) compared to healthy skin

SECONDARY OUTCOMES:
Comparison of visible scarring with the use of the CellutomeTM 12 months post baseline | 12 months
Comparison of impact of therapy on time to healing as assessed by ≥90% epithelialization 12 months post baseline. | 12 months
Comparison of chronic outcomes of therapy 12 months post baseline | 12 Months
  Assessed by the following: Vancouver Scar Scale (Vascularity 0-3; Pigmentation 0-3; Pliability 0-5; and Height 0-4)
Comparison of chronic outcomes of therapy 12 months post baseline | 12 Months
  Patient Observer Scar Assessment Scale (POSAS - evaluating patient perception of the scar including pain; itching; color; stiffness; thickness; irregularity on a 1-10 Likert Scale)
Comparison of chronic outcomes of therapy 12 months post baseline | 12 Months
  Visual assessment of Erythema of the donor site as compared to healthy skin
Comparison of chronic outcomes of therapy 12 months post baseline | 12 Months
  Visual assessment of Pigmentation of the donor site as compared to healthy skin
Comparison of chronic outcomes of therapy 12 months post baseline | 12 Months
  Elasticity of the donor site (measured with cutometer) compared to healthy skin.
Comparison of chronic outcomes of therapy 12 months post baseline | 12 Months
  Thickness (measured with ultrasound) compared to healthy skin
Comparison of chronic outcomes of therapy 12 months post baseline | 12 Months
  Sensation (measured by Semmes-Weinstein) compared to healthy skin

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid Blome-Eberwein, MD, Principal Investigator — Lehigh Valley Health Network
Locations (1):
- Lehigh Valley Health Network, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No